CLINICAL TRIAL: NCT05412693
Title: Six Weeks Functional Orthosis Versus Cast Immobilization for Partially Unstable Weber B/SER4a Ankle Fractures - a Multicenter Randomized Non-inferiority Trial
Brief Title: Functional Orthosis Versus Cast Immobilization for Partially Unstable Weber B Ankle Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: Alesund Hospital (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Marius Molund, Head of Foot and Ankle Service, Ostfold Hospital Trust
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22/00257-3
Record Dates: First submitted 2022-05-06; First posted 2022-06-09 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Ankle Fractures
Keywords: Weber B; SER4a
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking is not possible during the first 6 weeks of treatment due to the nature of the interventions. Investigators and outcome assessors will be masked for follow-up after 6 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional orthosis (Experimental): Use of a functional orthosis device (AirCast Air-Stirrup) for 6 weeks. Weightbearing as tolerated will be allowed in both groups immediately after application of the cast or orthosis.
  Interventions: Device: Functional orthosis
- Cast immobilization (Active Comparator): Use of a below-the-knee cast circular cast (3M scotch cast) for 6 weeks.
  Interventions: Device: Cast immobilization

INTERVENTIONS:
Device: Functional orthosis — See arm descriptions
  Arms: Functional orthosis
Device: Cast immobilization — See arm descriptions
  Arms: Cast immobilization

SUMMARY:
Stability dictates treatment choice for trans-syndesmotic fibula fractures. Optimal treatment for partially unstable fractures remains a topic of debate. The purpose of this study is to evaluate possible outcome non-inferior of functional orthosis treatment versus cast immobilization for these fractures.

DETAILED DESCRIPTION:
Evidence suggests that Weber B ankle fractures should be treated nonoperatively if the ankle mortise is stable. Stability is maintained if the deltoid ligament is intact, also known as a Weber B/SER2 injury. Functional orthosis treatment is advised for these injuries. Recently, authors have demonstrated that the fractured ankle can be functionally stable even with a partial deltoid ligament injury. Our interpretation of a partial deltoid ligament injury is when weightbearing radiographs indicate stability (no increase in medial clear space), while concomitant gravity stress radiographs indicate instability (due to increase in medial clear space). It is suggested that this is referred to as a Weber B/SER4a injury. Although now considered for nonoperative treatment, partially unstable/SER4a injuries were traditionally treated operatively. Today, the superiority of one method of nonoperative treatment over another for partially unstable/SER4a injuries remains unclear. Some authors advocate cast immobilization while others have shown good outcomes after inconsistently using different orthoses and cast devices. The argument for cast immobilization appears to be a fear of posttraumatic osteoarthritis because of potential recurrent instability. As a result, cast immobilization of partially unstable/SER4a fractures is implemented in reference European guidelines, and thus must be considered the reference treatment. To our knowledge, no study has documented increased prevalence of osteoarthritis associated with functional treatment of partially unstable/SER4a fractures. The use of cast immobilization remains a precautionary principle, but the choice is not so clear cut because cast immobilization comes with an increased risk of joint stiffness and thromboembolic complications. Long-term radiographic and patient-reported outcome data evaluating possible non-inferiority of functional orthosis treatment compared to cast immobilization will assist in guiding future treatment strategies of these common fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients:
* With isolated Weber type B fractures that are deemed stable on weightbearing radiographs (MCS injured ankle - MCS uninjured ankle < 1 mm).
* With concomitant gravity stress test evaluated as unstable (MCS injured ankle - MCS uninjured ankle < 1 mm)
* Presenting to one of the participating hospitals, and that are available for stability evaluation within 14 days after injury.
* 18-80 years of age
* With pre-injury walking ability without aids.

Exclusion Criteria:

* Patients:
* with fracture of the medial malleolus, pre-hospital closed fracture reduction, open fracture, fracture resulting from high-energy trauma or multi-trauma or pathologic fracture.
* with fracture of the posterior malleolus involving 25% or more of the joint surface or with a step of the intraarticular surface. (non-displaced fractures smaller than 25% can be included)
* with neuropathies and generalized joint disease such as Rheumatoid Arthritis.
* that are assumed not compliant (drug use, cognitive- and/or psychiatric disorders).
* with previous history of ipsilateral ankle fracture.
* with previous history of ipsilateral major ankle-/foot surgery.
* who live outside one of the participating hospitals catchment areas (not available for follow-up).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Between-groups difference in Manchester-Oxford Foot and Ankle Questionnaire score at 2 years | 2 years
  Scale 0-100, lower scores indicate less pain and symptoms.

SECONDARY OUTCOMES:
Between-groups difference in Olerud Molander Ankle Score at 2 years | 2 years
  Scale 0-100, higher scores indicate less pain and symptoms.
Numeric rating scale of of patient satisfaction with treatment protocol | 6 weeks
  A 0-10 rating scale for perceived satisfaction with orthosis or cast
Tibiotalar congruity comparing injured and uninjured ankle at 2 years | 2 years
  Measurement of ankle medial clear space from weightbearing and gravity stress ankle radiographs
Registrations of complications/adverse events | 2 years
  Registration of possible loss of congruence, delayed union, non-union, thromboembolic events
Change from 6 weeks ankle range of motion at 2 years | 6 weeks, 2 years
  Measurement using a goniometer (ad modum Lindsjø)

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (3):
  - Ålesund Hospital, Ålesund
  - Sykehuset Innlandet, Gjøvik, Gjøvik
  - Østfold Hospital Trust, Sarpsborg, Østfold fylke

IPD SHARING:
Plan to Share IPD: No